CLINICAL TRIAL: NCT02863705
Title: A 12-Month, Phase 4, Open Label, Multicenter, Trial to Assess the Efficacy and Safety of COMBIGAN® in Korean Patients With Primary Open Angle Glaucoma (POAG) and Normal Tension Glaucoma (NTG)
Brief Title: Efficacy and Safety of COMBIGAN® in Korean Patients With Primary Open Angle Glaucoma (POAG) and Normal Tension Glaucoma (NTG)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO-AP-EYE-0428
Record Dates: First submitted 2016-05-02; First posted 2016-08-11 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Glaucoma, Open-Angle; Normal Tension Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma | interventions — Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMBIGAN® (Experimental): One drop of COMBIGAN® in the affected eye, administered twice daily for 12 months
  Interventions: Drug: brimonidine tartrate/timolol malate Ophthalmic Solution
- COMBIGAN® + LUMIGAN® 0.01% (Experimental): LUMIGAN® will be administered once daily in the evening 5 minutes after COMBIGAN® instillation in patients who require additional IOP lowering.
  Interventions: Drug: brimonidine tartrate/timolol malate Ophthalmic Solution; Drug: bimatoprost ophthalmic solution 0.01%

INTERVENTIONS:
Drug: brimonidine tartrate/timolol malate Ophthalmic Solution — One drop of brimonidine tartrate/timolol malate (COMBIGAN®) Ophthalmic Solution in the affected eye, administered twice daily for 12 months
Drug: bimatoprost ophthalmic solution 0.01% — Bimatoprost ophthalmic solution 0.01% (LUMIGAN®) administered once daily in the evening 5 minutes after COMBIGAN® instillation if additional lowering IOP is needed
  Arms: COMBIGAN® + LUMIGAN® 0.01%

SUMMARY:
The objective of this study is to evaluate the long-term efficacy and safety of COMBIGAN® (brimonidine tartrate/timolol malate) in patients only using COMBIGAN® (brimonidine tartrate/timolol malate) and also in patients who require additional IOP lowering with LUMIGAN® (bimatoprost) 0.01%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Primary open angle glaucoma (Regardless of Intraocular pressure)
* Previous history of topical beta-blocker use and insufficiently controlled IOP

Exclusion Criteria:

* Pigmentary or exfoliative glaucoma
* History of angle-closure or an occludable angle by gonioscopy
* Prior filtration or laser iridotomy
* Argon laser trabeculoplasty or Selective laser trabeculoplasty performed less than 6 months
* History or signs of chronic inflammatory eye disease, ocular trauma, or potentially progressive retinal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Mean IOP change from Baseline (11AM point) | Baseline, Month 12

SECONDARY OUTCOMES:
Mean IOP change from Baseline (11AM point) | Baseline, Month 12
  Mean IOP change from baseline (11AM point) in the following patient sub-groups
  1. patients with NTG
  2. patients with POAG
  3. patients taking Combigan alone
  4. patients taking Combigan plus additional Lumigan 0.01%
Mean IOP change from Baseline (9AM point) | Baseline, Month 12
  Mean IOP change from baseline (9AM point) in the following patient sub-groups
  1. patients with NTG
  2. patients with POAG
  3. patients taking Combigan alone
  4. patients taking Combigan plus additional Lumigan 0.01%
Mean change in Mean deviation (MD) from Baseline | Baseline, Month 12
Mean change in Pattern standard deviation (PSD) from Baseline | Baseline, Month 12
Mean change in Visual field index (VFI) from Baseline | Baseline, Month 12
Mean change in cup to disc ratio (C/D ratio) from Baseline | Baseline, Month 12
Rate of VF progression measured as change in VF index over time | Baseline, Month 12
  Rate of VF progression during 12 months in the following patient sub-groups.
  1. patients with NTG
  2. patients with POAG
  3. patients taking Combigan alone
  4. patients taking Combigan plus additional Lumigan 0.01%
Mean duration of achieving the target IOP with COMBIGAN® alone | 12 Months
The percentage of subjects of achieving the target IOP with COMBIGAN® alone during 12 months | 12 Months
Definition of patient demographics (descriptive analysis of age and gender) | Baseline, Month 12
  Define patient demographics in the following patient sub-groups:
  1. patients with NTG
  2. patients with POAG
  3. patients taking Combigan alone
  4. patients taking Combigan plus additional Lumigan 0.01%

CONTACTS AND LOCATIONS:
Overall Officials: Joy Maglambayan, Study Director — Allergan
Locations (9):
- South Korea (9):
  - Pusan National University Hospital, Pusan National University School of Medicine, Busan
  - Yeungnam University Hospital, Yeungnam University College of Medicine, Daegu
  - Chungnam National University Hospital, Chungnam National University College of Medicine, Daejeon
  - Chonnam National University Hospital, Chonnam National University Medical School, Gwangju
  - Seoul National University Bundang Hospital, Seoul National University College of Medicine, Gyeonggi-do
  - Seoul National University Hospital, Seoul National University College of Medicine, Seoul
  - Kangbuk Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea College of Medicine, Seoul
  - Kim's Eye Hospital, Konyang University College of Medicine, Seoul